CLINICAL TRIAL: NCT05021354
Title: Effectiveness Of A Physiotherapy Treatment Plan In Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23/08/2021
Record Dates: First submitted 2021-08-23; First posted 2021-08-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Humeral Epicondylitis, Lateral
Keywords: Dry needling; Stretching; Eccentric exercise; tennis elbow; humeral epicondylitis, lateral
MeSH Terms: conditions — Tennis Elbow | interventions — Dry Needling; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling+eccentric exercises (Experimental): It is established a plan of treatment base on the evidence for dry needling, eccentric exercise in the patient with lateral epicondylalgia. This is done in two sessions, one session every 10 days and with a duration of about 45 minutes.
  Interventions: Device: Dry needling
- topical gel (Active Comparator): application of topical gel to the area of pain
  Interventions: Device: Topical gel
- NSAIDs (Active Comparator): oral intake of NSAIDs
  Interventions: Drug: NSAIDs

INTERVENTIONS:
Device: Dry needling — dry needling, stretching and eccentric exercise
  Arms: Dry needling+eccentric exercises
Device: Topical gel — aplication of topical gel to the epicondyle
  Arms: topical gel
Drug: NSAIDs — oral intake of NSAIDs
  Arms: NSAIDs

SUMMARY:
Purpose: Test the effectiveness of a physiotherapy treatment in 90 patients with Lateral epicondylalgia (LE).

DETAILED DESCRIPTION:
Methods: LE is a musculoskeletal pain around the lateral epicondyle that may also present with decreased grip strength and/or neuromuscular disorders. An evidence-based treatment plan of dry needling, stretching and eccentric exercise in the patient with lateral epicondylalgia is established. It is carried out in two sessions, one session every 10 days and lasts about 45 minutes. There are three intervention arms: dry needling, atopic gel and NSAIDs, 30 patients in each group (n=90).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with lateral epicondylalgia

Exclusion Criteria:

* diagnosed with compressive nerve syndromes with irradiation to the upper limb

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Questionaire Hand 10 | 1 month
  score in discomfort hand 0-10. 0 is the lowest score and 10 is the highest score.
VAS Scale | 1 month
  pain scale, where 0 is the minimum pain and 10 is the maximum pain.

SECONDARY OUTCOMES:
pain concentration measured with algometry | 10 days
  pain when performing static pressures measured with an algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heales LJ, Bergin MJG, Vicenzino B, Hodges PW. Forearm Muscle Activity in Lateral Epicondylalgia: A Systematic Review with Quantitative Analysis. Sports Med. 2016 Dec;46(12):1833-1845. doi: 10.1007/s40279-016-0539-4. PMID 27106557
- [Background] Aguilera-Eguía R, Ibacache-Palma A, Ignacia-Ulloa M, Flores-Fernández C, López-Soto LM, López Soto OP. Effectiveness of acupuncture in patients with lateral epicondylalgia: an overview of systematic reviews. Rev Cienc Salud. 2017;15(1):37-48.
- [Background] Araya Quintanilla F, Moyano Galvez V. Exercise therapy for lateral epicondylalgia: Systematic review. Rev Soc Esp Dolor 2015;22(6):253-270.
- [Background] Aguilera Eguía RA, Zafra Santos EO, Rojas López DK, Saavedra Rozas PA, Cofre Bolados C. Effectiveness of low frequency laser in the treatment of pain in patients with lateral epicondylalgia: An overview of systematic reviews. Rev Soc Esp Dolor 2015; 22(1): 39-47.
- [Background] Patel RM, Lynch TS, Amin NH, Calabrese G, Gryzlo SM, Schickendantz MS. The thrower's elbow. Orthop Clin North Am. 2014 Jul;45(3):355-76. doi: 10.1016/j.ocl.2014.03.007. PMID 24975763
- [Background] Dones VC 3rd, Grimmer K, Thoirs K, Suarez CG, Luker J. The diagnostic validity of musculoskeletal ultrasound in lateral epicondylalgia: a systematic review. BMC Med Imaging. 2014 Mar 3;14:10. doi: 10.1186/1471-2342-14-10. PMID 24589069
- [Background] Cha YK, Kim SJ, Park NH, Kim JY, Kim JH, Park JY. Magnetic resonance imaging of patients with lateral epicondylitis: Relationship between pain and severity of imaging features in elbow joints. Acta Orthop Traumatol Turc. 2019 Sep;53(5):366-371. doi: 10.1016/j.aott.2019.04.006. Epub 2019 Apr 28. PMID 31040053
- [Background] Lee JH, Kim TH, Lim KB. Effects of eccentric control exercise for wrist extensor and shoulder stabilization exercise on the pain and functions of tennis elbow. J Phys Ther Sci. 2018 Apr;30(4):590-594. doi: 10.1589/jpts.30.590. Epub 2018 Apr 20. PMID 29706713
- [Result] Bisset LM, Vicenzino B. Physiotherapy management of lateral epicondylalgia. J Physiother. 2015 Oct;61(4):174-81. doi: 10.1016/j.jphys.2015.07.015. Epub 2015 Sep 8. No abstract available. PMID 26361816
- [Result] George CE, Heales LJ, Stanton R, Wintour SA, Kean CO. Sticking to the facts: A systematic review of the effects of therapeutic tape in lateral epicondylalgia. Phys Ther Sport. 2019 Nov;40:117-127. doi: 10.1016/j.ptsp.2019.08.011. Epub 2019 Aug 27. PMID 31518778
- [Result] Dong W, Goost H, Lin XB, Burger C, Paul C, Wang ZL, Kong FL, Welle K, Jiang ZC, Kabir K. Injection therapies for lateral epicondylalgia: a systematic review and Bayesian network meta-analysis. Br J Sports Med. 2016 Aug;50(15):900-8. doi: 10.1136/bjsports-2014-094387. Epub 2015 Sep 21. PMID 26392595
- [Result] Nishizuka T, Iwatsuki K, Kurimoto S, Yamamoto M, Onishi T, Hirata H. Favorable Responsiveness of the Hand10 Questionnaire to Assess Treatment Outcomes for Lateral Epicondylitis. J Hand Surg Asian Pac Vol. 2018 Jun;23(2):205-209. doi: 10.1142/S2424835518500212. PMID 29734897
- [Result] Uygur E, Aktas B, Ozkut A, Erinc S, Yilmazoglu EG. Dry needling in lateral epicondylitis: a prospective controlled study. Int Orthop. 2017 Nov;41(11):2321-2325. doi: 10.1007/s00264-017-3604-1. Epub 2017 Aug 21. PMID 28828509
- [Derived] Sanchez-Mila Z, Abuin-Porras V, Fidalgo-Gomez H, Minguez-Esteban I, Almazan-Polo J, Velazquez-Saornil J. Efficacy of Dry Needling Combined with Eccentric Exercise Versus Oral and Topical NSAID Treatment in Patients with Tennis Elbow: A Randomized Controlled Trial. J Evid Based Integr Med. 2025 Jan-Dec;30:2515690X251355017. doi: 10.1177/2515690X251355017. Epub 2025 Jul 9. PMID 40629912